CLINICAL TRIAL: NCT04611945
Title: Westlake Sailing Cohort: Dynamic Change of Human Microbiome During Sailing
Brief Title: Westlake Sailing Cohort
Status: Completed | Type: Observational
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Other Study IDs: 20200911ZJS001
Record Dates: First submitted 2020-10-09; First posted 2020-11-02 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Microbiome; Glucose Metabolism; Mood; Environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, white cells, urine, faeces, tongue coating, skin microbiome
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Little is known about the dynamic change of human microbiome in different body sites including skin, mouth and gut during sailing. The present study aims to reveal the change of human microbiome in response to the sailing environment in a 1-month period, and its implication for human health.

DETAILED DESCRIPTION:
This study will recruit a number of participants who are going to sail for mariana trench from Shenzhen, China. Characteristics of the participants will be described by a series of index of stool, urine, skin microbiota and tongue coating. All the biospecimen will be collected before and during the voyage. Stool at the 2nd, the 4th and the 12th week after the voyage and blood sample at the baseline will also be collected. Participants' mood states, health-related quality of life, fatigue score and sleep quality will be investigated with questionnaires throughout the 1-month period. Participants are asked to record diseases and symptoms, if any, when sailing. All the data will be used to analyse how microbiota change and be involved in human health during a voyage.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and capability to complete the study protocol

Exclusion Criteria:

* Inability or unwillingness to approved to provide informed consent.
* Women who are pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who will sail by Shenkuo, a scientific research ship, December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Gut microbial abundant change | Day 1, day 10, day 16, day 23, day 28
  Gut microbial communities and their abundant features will be analysed based on shotgun metagenomic sequencing.
Tongue coating microbial abundant change | Day 1, day 10, day 16, day 23, day 28
  Tongue coating microbial communities and their abundant features will be analysed based on shotgun metagenomic sequencing.

SECONDARY OUTCOMES:
Mood states change over 4 weeks | Day 1, day 10, day 16, day 23, day 30
  Transient, fluctuating feelings, and enduring affect states will be assessed by the Profile of Mood States-Short Form (POMS-SF) . POMS-SF contains 30 questions that assess the following seven different moods: anger-hostility (AH), confusion-bewilderment (CB), depression-dejection (DD), fatigue-inertia (FI), tension-anxiety (TA), vigoractivity (VA), and friendliness (F). Total mood disturbance (TMD) scores were calculated based on the previous seven factors. High scores for VA and F indicate a positive mood state, while high scores for AH, CB, DD, FI, TA, and TMD indicate a negative mood state.
Health-related quality of life change over the one-month sailing | Day 1, day 30
  Health-related quality of life will be assessed by the Short-Form 36 Health Status Questionnaire（SF-36). It contains eight subscales scoring from 0 to 100 points for each, with higher scores indicating better quality of life.
Sleep quality change over the one-month sailing | Day 1, day 30
  The Pittsburgh Sleep Quality Index （PSQI）will be used to assess sleep quality. It comprises 19 items for self-reported sleep quality in the last month and five additional questions to be answered by roommates, if applicable. The 19 items are grouped into seven component scores: sleep quality, sleep latency, sleep duration, efficiency of habitual sleep, sleep disturbance, use of sleep medication, and diurnal dysfunction. These are then added to a global PSQI score. The PSQI score ranges from 0 to 21, with a higher score indicative of poorer sleep quality.
Short-chain fatty acids change | Day 1, day 10, day 16, day 23, day 28
  Short-chain fatty acids will be analysed by performing liquid chromatography/quadrupole time-of-flight mass spectrometry (LC/Q-TOF/MS).
Weight change | Day 1, day 10, day 16, day 23, day 28
  Weight will be described by kilogram.
Blood pressure change | Day 1, day 10, day 16, day 23, day 28
  Systolic pressure and diastolic pressure will be measured and described by mmHg.
Fatigue score change | Day 1, day 10, day 16, day 23, day 30
  The Multi-dimensional Fatigue Inventory (MFI-20) will be used to measure aspects of fatigue experienced during the previous days. It consists of five subscales of fatigue: general fatigue (GF), physical fatigue (PF), re-duced motivation (RM), reduced activity (RA), and mental fatigue (MF). The score ranges from 20 to 100. Higher scores indicate a higher degree of fatigue.
Skin microbial abundant change | Day 1, day 10, day 16, day 23, day 28
  Skin microbial communities and their abundant features will be analysed based on shotgun metagenomic sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, Principal Investigator — Westlake University
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided